CLINICAL TRIAL: NCT02481843
Title: Hyperoxia, Erythropoiesis and Tissue Oxygenation in Critically Ill Patient
Brief Title: Hyperoxia, Erythropoiesis and Microcirculation in Critically Ill Patient
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Associate Professor and Medical Doctor, Università Politecnica delle Marche
Other Study IDs: NOP001
Record Dates: First submitted 2015-06-15; First posted 2015-06-25 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Failure
Keywords: Hyperoxia; Microcirculation; Erythropoietin; Normobaric Oxygen Paradox
MeSH Terms: conditions — Respiratory Insufficiency; Hyperoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hyperoxia: 2-hours of hyperoxia (FiO2 = 1.0)
  Interventions: Other: 2 hours of hyperoxia (FiO2 = 1)
- Control: 2-hours control without hyperoxia

INTERVENTIONS:
Other: 2 hours of hyperoxia (FiO2 = 1) — Patients received 2 hours of hyperoxia at FiO2 = 1
  Other Names: Hyperoxia
  Groups: Hyperoxia

SUMMARY:
Prospective observational study in 40 adult critically ill patients. Patients were eligible if they were mechanically ventilated with an FiO2 ≤0.5 and PaO2/FiO2 ≥200 mmHg and hemodynamically stable with a hemoglobin ≥9 g/dL, no acute bleeding or need for blood transfusions, no renal failure, no chronic obstructive pulmonary disease. Twenty patients (hyperoxia group) underwent a 2-hour exposure to normobaric hyperoxia (FiO2 1.0), 20 patients were evaluated as controls. Serum erythropoietin (EPO) was measured at baseline, 24h and 48h. Serum Glutathione (GSH) and reacting oxygen species (ROS) were assessed at baseline (t0), after 2 hours of hyperoxia (t1) and 2 hours after the return to baseline FiO2 (t2). Sidestream dark field videomicroscopy was applied sublingually to assess the microvascular response to hyperoxia. Near infrared spectroscopy with a vascular occlusion test was applied at t0, t1, t2.

DETAILED DESCRIPTION:
Interventions:

Forty patients were enrolled in total. The first 20 patients (hyperoxia group) underwent a 2-hour period of normobaric hyperoxia (FiO2 1.0), according to the protocol applied in. No variation in the FiO2 was applied for the other 20 patients (control group). All patients were enrolled in the morning and hyperoxia was performed in the time range between 10am-2pm in order to minimize variability due to the circadian rhythm of EPO production. No variations to sedation or vasopressor dose were applied during the study period.

Measurements:

On the study day, measurements were taken at 2-hour intervals: baseline (t0), under 1.0 FiO2 (t1) and after returning to baseline FiO2 (t2). These included: body temperature, heart rate (HR), mean arterial pressure (MAP), arterial oxygen saturation (SaO2), arterial partial pressure of oxygen (PaO2) and carbon dioxide (PaCO2), PaO2/FiO2, arterial pH, bicarbonate, base excess) and central venous saturation (ScvO2) blood gases, arterial lactates, evaluation of the sublingual microcirculation and tissue oxygenation. The same measurements were performed in the control group at 2-hour intervals. In 24 patients (12 patients per group), arterial blood samples (10 mL) were taken at each time point and immediately centrifuged; plasma and serum were stored at -70°C for subsequent analyses. Serum EPO, reticulocyte count, hemoglobin (Hb) and hematocrit were measured at 8am in all patients on the study day, at 24 and 48 hours.

Microcirculation measurements with sidestream dark field imaging The sublingual microcirculation was evaluated with sidestream dark field (SDF) videomicroscopy (Microscan, Microvision Medical, Amsterdam, NL). This technique has been described in details elsewhere.

Poor-quality images were discarded, and three images for each time point were selected and analyzed by using a computer software package (Automated Vascular Analysis Software; Microvision Medical BV). According to the consensus report on the performance and evaluation of microcirculation using SDF imaging, total vessel density (TVD), perfused vessel density (PVD), De Backer score, proportion of perfused vessels (PPV), microcirculatory flow index (MFI), flow heterogeneity index (FHI) and blood flow velocity (BFV) were calculated in small or medium vessels (diameter ≤ or >20 μm, respectively), as previously described. In addition to discontinuous microvascular measurements at 2-hour intervals, the investigators evaluated the early response of the microcirculation to variations in the FiO2 on one and the same site of sublingual mucosa in order to detect even minute changes in the microvascular density and flow. Directly after obtaining measurements from 5 different sites, the SDF probe was placed in a stable position and manipulated to avoid any pressure artifacts or secretions interfering with the analysis. By manually supporting the microscope, continuous video recording was performed for at least 2 minutes during the variation of the FiO2 (start or end of hyperoxia). Video clips of 10 s (2 per time point) corresponding to before (baseline or 2h FiO2 1.0) and after (2 min FiO2 1.0 or 2 min after returning to baseline FiO2) the variation of FiO2 were subsequently selected and analyzed.

Evaluation of peripheral tissue oxygenation and microvascular reactivity with near infrared spectroscopy.

Near-infrared reflectance spectrophotometry (NIRS) (InSpectra™ Model 650; Hutchinson Technology Inc., Hutchinson, USA) was used to measure peripheral tissue oxygen saturation (StO2) and tissue Hb index (THI) at baseline and during a vascular occlusion test (VOT). A 15 mm-sized probe was placed on the skin of the thenar eminence, and a sphygmomanometer cuff was placed around the (upper) arm to occlude the brachial artery. After a 3-minute period of StO2 signal stabilization, arterial inflow was arrested by inflation of the cuff to 50 mmHg above the systolic arterial pressure. The cuff was kept inflated until the StO2 decreased to 40% and then released. StO2 was continuously recorded during the reperfusion phase until stabilization. The StO2 downslope (%/minute) was calculated from the regression line of the first minute of StO2 decay after occlusion, providing an index of O2 consumption rate. The StO2 upslope (%/minute) was obtained from the regression line of StO2 increase in the reperfusion phase. The area under the curve (AUC) of the hyperemic response was also calculated. StO2 upslope and the AUC of the StO2 reflect microvascular reactivity. All the parameters were calculated by using a computer software package (version 3.03 InSpectra Analysis Program; Hutchinson Technology Inc.).

Immunoassays :

Levels of ROS and GSH were measured in accordance with the instructions of the manufacturer.

Statistical analysis:

Statistical analysis was performed by using GraphPad Prism version 6 (GraphPad Software, USA). Normality of distribution was checked by using the Kolmogorov-Smirnov test. Data were presented as mean ± standard deviation or median [1st-3rd quartile], as appropriate. One-way analysis of variance (ANOVA) for repeated measures with Bonferroni post-hoc test or Friedman test with Dunn's multiple comparison test were used to evaluate changes over time in the same group. Two-way ANOVA for repeated measures with Bonferroni post-hoc test was used to evaluate differences between the two groups, where applicable. For non-normally distributed variables, the Mann-Whitney U test was applied to evaluate difference between the two groups at the same time point. A Spearman correlation coefficient was calculated to assess correlations between variables. The alpha level of significance was set a priori at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical Ventilated Patients

Exclusion Criteria:

* PaO2/FiO2 < 200
* hemoglobin (Hb) <9 g/dL
* acute bleeding or blood transfusions during the study period
* any surgical interventions during the study period
* acute or chronic renal failure
* hemodynamic instability
* chronic obstructive pulmonary disease
* pregnancy
* factors impeding the sublingual microcirculation evaluation (oral surgery or facial trauma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18-year old) patients admitted to a 12-bed medical-surgical ICU
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Normobaric Oxygen Hyperoxia in increasing serum erythropoietin levels in critically ill patients | up to 2 day after FiO2=1 exposure
  Blood samples to detect erythropoietin

SECONDARY OUTCOMES:
Effects of hyperoxia on the sublingual microcirculation | Before FiO2, after 2 hours of FiO2=1 exposure, 2 hours after the end of FiO2=1 exposure
  SDF technique will be used to look at sublingual microcirculation, 20 seconds movies are registered and software is used to analyze them
Effects of hyperoxia on the peripheral microcirculation | Before FiO2 = 1, after 2 hours of FiO2=1 exposure, 2 hours after the end of FiO2=1 exposure
  Near Infra-Red Spectroscopy is used to assess oxygen tissue saturation at thenar and vascular occlusion test is performed to assess the desaturation and resaturation curves
Hyperoxia and variations in circulating glutathione | Before FiO2 = 1, after 2 hours of FiO2=1 exposure, 2 hours after the end of FiO2=1 exposure
  Blood samples
Hyperoxia and variations in circulating nitric oxide | Before FiO2 = 1, after 2 hours of FiO2=1 exposure, 2 hours after the end of FiO2=1 exposure
  Blood samples
Hyperoxia and variations in circulating ROS | Before FiO2 = 1, after 2 hours of FiO2=1 exposure, 2 hours after the end of FiO2=1 exposure
  Blood samples
Reticulocyte Count | Before FiO2 = 1, at 1 day and 2 day after FiO2=1 exposure
Effectiveness of Normobaric Oxygen Hyperoxia in increasing serum erythropoietin levels in critically ill patients after 1 day | Before FIO2 = 1 and at 1 day after FiO2 = 1 exposure

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, Principal Investigator — AOU Ospedali Riuniti Ancona
Locations (1):
- University ICU, AOU Ospedali Riuniti Ancona, Torrette Di Ancona, Ancona, Italy

REFERENCES:
- [Derived] Donati A, Damiani E, Zuccari S, Domizi R, Scorcella C, Girardis M, Giulietti A, Vignini A, Adrario E, Romano R, Mazzanti L, Pelaia P, Singer M. Effects of short-term hyperoxia on erythropoietin levels and microcirculation in critically Ill patients: a prospective observational pilot study. BMC Anesthesiol. 2017 Mar 23;17(1):49. doi: 10.1186/s12871-017-0342-2. PMID 28335733